CLINICAL TRIAL: NCT03777800
Title: Body Therapy for War Veterans With Post Traumatic Stress Disorder (PTSD): A Combined Randomized Controlled Trial (RCT) and Qualitative Study.
Brief Title: Body Therapy for War Veterans With Post Traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: National Board of Health, Denmark (Other Government); Soldaterlegatet (Unknown); ManuVision (Unknown); Copenhagen University Hospital, Denmark (Other); Patientforeningen Danmark (Unknown)
Responsible Party: Principal Investigator, Susan Andersen, Principal investigator, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10.128
Record Dates: First submitted 2018-12-11; First posted 2018-12-17 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Stress Disorders, Post-Traumatic; Trauma and Stressor Related Disorders; Behavioral Symptoms; Depression; Quality of Life
Keywords: Veterans; Nervous System Diseases; Body Therapy; Mind-Body Therapies; Coping Skills; Breathing techniques; Body awareness; Emotional regulation; Randomized Controlled Trial; Qualitative study; Mixed-methods
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Trauma and Stressor Related Disorders; Behavioral Symptoms; Depression; Nervous System Diseases; Emotional Regulation | interventions — Mind-Body Therapies; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Body Therapy (Experimental): Participants in the intervention condition will be assigned to a 6-month body therapy treatment focused on 24 individual body treatments including conversations and direct physical treatment of the body combined with home-based daily practice of meditation.
  Interventions: Behavioral: Body therapy
- Treatment As usual (Active Comparator): Participants in the control condition will be offered treatment as usual, which is psychiatric medication and/or individual psychotherapy as deemed relevant by the psychiatrist.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Body therapy — Body therapy involving direct physical treatments, conversations, breathing exercises and relaxation in the sessions. Moreover, the participants are taught how to practice vipassana or awareness meditation every day at home.
  The body therapist works directly with the muscle armour and the treatment sessions have focus on creating a safe environment and enabling cognitive realisation and awareness of symptoms.
  Each participant is assigned a practitioner who acts as contact person and 'lifeline'. Furthermore, a coordinator is assigned in ManuVision who will also act as contact person when needed for the veterans. This provides peace of mind, trust, and ensures retention. The coordinator or the practitioner follows up on the veteran's progress prior to each session.
  Other Names: ManuVision
  Arms: Body Therapy
Behavioral: Treatment as usual — Standard treatment
  Arms: Treatment As usual

SUMMARY:
The present study is a randomized, controlled trial that compares a certain type of body therapy, called ManuVision, to treatment as usual (TAU) in war veterans with posttraumatic stress disorder (PTSD). The purpose of the study is to determine whether participation in the body therapy treatment by war veterans who have PTSD, will reduce symptoms of PTSD and depression, and improve quality of life, function level and body awareness.

Study hypotheses state that the ManuVision approach, compared to the treatment as usual, will be more effective at reducing the PTSD symptoms experienced by veterans because it will help the veterans learning to become aware of, accept the PTSD symptoms, reading their own emotional state and gain body awareness and subsequently have emotional control and improved coping mechanism when PTSD symptoms arise. The awareness, accept and improved coping mechanisms means that the nervous system is not under the same pressure and that PTSD symptoms therefore may be reduced.

DETAILED DESCRIPTION:
Background: A sizable proportion of soldiers involved in military missions are experiencing mental health and adjustment problems on their return, including PTSD. PTSD is both a psychological and a physical condition, which occurs as a post-reaction to one or more traumatic experiences. The symptoms include aggressive behaviour, difficulty sleeping, tiredness, anxiety, and social isolation, and many sufferers develop depression, and the war veterans are at a higher risk of suicide. Physiologically, people with PTSD experience an activation of their sympathetic nervous system, whereby the stress hormones adrenalin and cortisol are released, the heart rate increases, the blood pressure rises, and the body is geared toward a 'fight or flight' response. A major challenge for veterans with PTSD is emotional control and problems with reading their own and others' emotional state.

This study will provide a certain type of body therapy, called ManuVision, to war veterans with PTSD. ManuVision is a Danish developed body therapy working with direct physical treatment of the body and through this approach with the client's psychosocial resources. There are conversations during and before treatment, as appropriate, and trust is intentionally built from the first meeting through eye contact and open breathing on behalf of the ManuVision therapist. The treatment is based on the understanding that chock, trauma and stress are stored in the body blocking the muscles and breathing and affecting the nerve system.

The intervention in this project entails individual courses of body therapy including 24 treatment sessions over 6 months for veterans with PTSD, plus recommended daily meditation at home.

The study goals are to:

1. Investigate how the body therapy treatment is implemented, and how the participants experience the treatment, respond to the treatment and which transformations participants experience in the everyday life (a process evaluation by qualitative methods).
2. Compare the body therapy treatment with treatment as usual (TAU). Symptoms of PTSD, depression, function level, quality of life, and body awareness will be examined at pre-treatment, midway during the treatment period, post-treatment and, if possible, at follow-up to determine if symptoms change over time (an effect evaluation by quantitative methods).

The research questions are as follows:

A. How is the treatment implemented, how do the participants experience and respond to the treatment, and what characterizes the interaction between veteran and practitioner? B. In which ways do the veterans experience transformations, e.g. in terms of their body, feelings, social relations, everyday lives, quality of life, and handling their PTSD symptoms? C. What is the effect of the intervention on PTSD symptoms, quality of life, function level, depression and body awareness? D. Are there better outcomes for participants who received more treatment (i.e., number of treatment sessions)?

In order to answer the research questions A and B we will use participant observation, qualitative interviews, and focus group interviews with veterans, family members and practitioners.

In order to answer the research question C concerning the intervention's effect, appropriate statistical methods (e.g., Repeated measures ANOVA) will be used to analyse the differences between the intervention and the control group based on validated questionnaires.

Finally, a dose-response analysis is carried out (D) based on the practitioners' registered number of treatment sessions. This will support and refine the effect estimations.

ELIGIBILITY:
Inclusion Criteria:

* Veterans
* Meet criteria for clinical PTSD or subclinical PTSD assessed by The Structured Clinical Interview for DSM-IV (SCID)
* Demonstrate understanding of informed consent and normal cognitive skills

Exclusion Criteria:

* Current substance dependence (alcohol or drugs)
* Severe mental disorders such as schizophrenia, Bipolar I or II disorder, or current psychiatric conditions such as psychosis or mania

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Self-reported PTSD symptoms by the PTSD checklist - military version (PCL-M) | Change from baseline to midway (approximately 3 months), post-treatment (approximately 6 months) and, if possible, follow-up (12 months)
  The PTSD checklist contains 17 items corresponding to the DSM-IV criteria for PTSD. Past month symptom severity is indicated using a 5 point scale. Higher scores represent greater severity.

SECONDARY OUTCOMES:
Self-reported depression symptoms as measured by the Major Depression Inventory (MDI) | Change from baseline to midway (approximately 3 months), post-treatment (approximately 6 months) and, if possible, follow-up (12 months)
  The severity of depression is measured over the last 2 weeks in the form of a Likert scale at which the frequency of each symptom can be indicated from 0 (at no time) to 5 (all the time). Score range is from 0 (no depression) to 50 (extreme depression).
Self-reported quality of life using the World Health Organization Five Well-Being Index (WHO-5) | Change from baseline to midway (approximately 3 months), post-treatment (approximately 6 months) and, if possible, follow-up (12 months)
  Each of the five items indicates current positive wellbeing during the previous two weeks from 0 (at no time) to 5 (all of the time).
Function level using the Sheehan Disability Scale (SDS) | Change from baseline to midway (approximately 3 months), post-treatment (approximately 6 months) and, if possible, follow-up (12 months)
  A self-administered rating scale measuring functional impairment with regard to family, work and social network using three visual analogue scales.
Self-reported body awareness using the Multidimensional Assessment of Interceptive Awareness (MAIA) Questionnaire | Change from baseline to midway (approximately 3 months), post-treatment (approximately 6 months) and, if possible, follow-up (12 months)
  MAIA contains 32 items. The items are organized into eight subscales: (1) Noticing: the awareness of body sensations; (2) Not-Distracting: the tendency to ignore or distract oneself from sensations of pain or discomfort; (3) Not-Worrying: emotional distress or worry with sensations of pain or discomfort; (4) Attention Regulation: the ability to sustain and control attention to body sensation; (5) Emotional Awareness: the awareness of the connection between body sensations and emotional states; (6) Self-Regulation: the ability to regulate psychological distress by attention to body sensations; (7) Body Listening: actively listening to the body for insight; (8) Trusting: experiencing one's body as safe and trustworthy.

OTHER OUTCOMES:
Participants' responsiveness | Post-treatment (approximately 6 months)
  A 3-item questionnaire with a 0-10 response scale to measure the participants' judgement of the treatment (only the intervention group)

CONTACTS AND LOCATIONS:
Overall Officials: Nanna Ahlmark, PhD, Principal Investigator — National Institute of Public Health, University of Southern Denmark
Locations (1):
- Military Psychiatric Center, Copenhagen University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ahlmark NG, Dahl A, Andersen HS, Tjornhoj-Thomsen T, Andersen S. Body therapy versus treatment as usual among Danish veterans with PTSD: Study protocol for a randomised controlled trial combined with a qualitative study. Contemp Clin Trials Commun. 2020 Jun 20;19:100596. doi: 10.1016/j.conctc.2020.100596. eCollection 2020 Sep. PMID 32617435